CLINICAL TRIAL: NCT03335462
Title: The Spread of Paravertebral Injections in the Lumbar Plexus Area and Associated Risk Factors to Adjacent Organs: a CT Scan Based Report
Brief Title: Spread of Paravertebral Injections in the Lumbar Plexus Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12112008
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Lumbar Plexus Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paravertebral injections (Experimental): Lumbar paravertebral injections containing contrast will be performed. The needles are kept in their position and afterwards followed by CT scan.
  Interventions: Other: Paravertebral injections; Other: CT scan

INTERVENTIONS:
Other: Paravertebral injections — Paravertebral injections will be performed in the thoraco-lumbar plexus area under CT guidance
Other: CT scan — CT scan will be performed as the needles are kept in their position after injecting the contrast

SUMMARY:
Lumbar paravertebral block (LPB) has been used for anesthesia in different settings such as in varicocelectomy and inguinal hernia repair in adults and pediatrics. Different studies considered LPB as an alternative to general and spinal anesthesia when contraindications exist, especially in elderly patients. However, the results obtained when using LPB are controversial in terms of number of injections performed and the success rates.

DETAILED DESCRIPTION:
Patients scheduled for hernia repair who will agree to undergo different number of paravertebral injections in the thoraco-lumbar plexus area under CT guidance.

While the patient is in lateral decubitis position, LPB injections will be made using a 100 mm 22 G nerve stimulator needle (Stimuplex, B.Braun, Melsungen, Germany). The site of injection is determined by manual palpation. The number of injections ranges from one to five and the level of injections ranges from T11 to L3.

The needle is penetrated perpendicular to the skin using the following nerve stimulator settings: 5mA, 9V and 2Hz. The stimulating needle is gently manipulated into a position to allow an adequate muscular response with a stimulating current of 0.4-0.8 mA. At this point, 4-5 ml of the contrast (Telebrix 35, 350 mg/ml, Roissy CDG Cedex, France) is injected. The patients will receive the same amount of contrast, despite the different number of injections. The needles are kept in their position and afterwards followed by CT scan.

A radiologist who is blind to the study will interpret the radiological results and document the level at which the needle tip is found, the distance from the kidney and the spread of the injected contrast. In order to ensure patient's safety, different measures will be taken to keep the radiation as low as reasonably achievable.

Following the radiological practice, patients will be transferred to the operating room to undergo inguinal herniorrhaphy, and will not followed for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Scheduled for hernia repair

Exclusion Criteria:

Patients

* with coagulation disorders,
* with infection at the injection site,
* with allergy to contrast
* receiving opioids

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Injection spread | 5 minutes after the procedure
  Demonstrate spread of injected material in the lumbar plexus area according to different number of injections confirmed by CT guidance

SECONDARY OUTCOMES:
Distance between injections and kidney | 5 minutes after the procedure
  Measure the distance between the injections and kidney to assess safety of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon